CLINICAL TRIAL: NCT04424108
Title: The Effect of Hormone Therapy on Serum Ischemia Modified Albumin Levels in Surgical Menopausal Women
Brief Title: Hormone Therapy on Serum Ischemia Modified Albumin in Menopausal Women
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, professor, Karadeniz Technical University
Other Study IDs: 2009/54
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Hormone Therapy Induced Morphologic Change; Surgical Menopause
Keywords: IMA; menopause; hormone therapy; cardiovascular risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Women suffer from cardiovascular diseases 10 years later than men, therefore female sex has been considered as a 'protective factor'. However, the risk of cardiovascular disease in women increases rapidly after menopause and the declining levels of endogenous estrogen is thought to be the causative factor. Furthermore, Postmenopausal hormone therapy (HT) decreases the severity and intensity of menopausal symptoms and improves women's quality of life. Until the last 10 years, based on the results of observational studies, postmenopausal HT may protect women against cardiovascular events and decrease the risk of coronary artery disease by 35-50%. However, recent randomized primary and secondary prevention trials did not support the cardioprotective effect of HT.

The aim of this study is to assess the effect of hormone therapy on serum ischemia modified albumin (IMA) levels. Thirty surgical menopausal women who admitted to Karadeniz Technical University, Faculty of Medicine, Department of Obstetrics and Gynecology during 1-year period and diagnosed as menopause and planned to have hormone therapy for menopausal symptoms were enrolled for this prospective study. The serum İMA levels were recorded before and after (3 months, 6 months, 12 months later) hormone treatment (2 mg Estradiol Hemihidrat).

ELIGIBILITY:
Inclusion Criteria:

* accepting consent to participate in the trial and signing the form
* Surgical menopausal women aged 45-55 (having TAH + BSO for benign reasons)
* Presence of vasomotor or menopausal symptoms (moderate to severe);
* no systemic disease or infectious disease in the past 2 weeks
* Not taking any other hormone therapy or medication until postoperative 6th week;
* no contraindications for hormone therapy in routine menopause evaluation;
* Willingness to take hormone therapy
* No smoking.

Exclusion Criteria:

* Any systemic disease presence
* Smoking
* Contraindications for hormone therapy
* Failure to follow-up
* Inability to complete three months of hormone therapy
* quitting hormone therapy for other medical reasons during hormone therapy
* Cases reported as preinvasive and invasive genital tumors as a result of TAH + BSO
* Cases reported as suspicious findings in the mammography report

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The treatment of menopause and hormone happens only in female sex.
Study Population: Within 10 months of the study period, estradiol hemihydrate for all patients who underwent TAH + BSO for gynecology and obstetrics in our clinic and evaluated with the diagnosis of surgical menopause in the postoperative period (6th week) was prescribed. These cases were evaluated in terms of inclusion and exclusion criteria after they were determined to be volunteers to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2010-05-01 (Actual); Study Completion 2010-05-20 (Actual)

PRIMARY OUTCOMES:
Measuring serum ischemia-modified albumin (IMA) level | 12 months
  After collecting all blood, serums were re-dissolved, and serum IMA levels were checked. IMA level was evaluated by the rapid colorimetric method developed by Barr-Or as an absorbance unit. For IMA, the results were recorded in the spectrophotometer at appropriate wavelengths, and the results were recorded as absorbance units.
Hormone therapy usage | 12 months
  Estradiol hemihydrate containing preparation 12 boxes in all patients given 1 tablet per day (2 mg / day) was prescribed as. Patients were recommended to reapply at the 3rd, 6th, and 12th months of treatment following drug use.